CLINICAL TRIAL: NCT02195752
Title: Observational Study of Patient and Physician Experiences During Treatment of Pain With Compounded Pharmaceuticals
Brief Title: Lexington Observational Study of Treatment With Compounded Pain Creams
Acronym: TrackingCPC
Status: Terminated | Type: Observational
Why Stopped: Sponsor financial decision stemming from low recruitment
Sponsor: Lexington Independent Studies, LLC (Industry)
Collaborators: Palm Beach CRO (Unknown)
Responsible Party: Sponsor
Other Study IDs: LIS001
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain; Acute Pain
Keywords: Compounded pain cream; Ordinary care; Compounding; Topical treatment; Analgesia
MeSH Terms: conditions — Chronic Pain; Acute Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prescribed Compounded Pain Cream: The study is limited to patients who have been prescribed treatment with a topical compounded pain cream as a component of their ordinary care by a qualified physician.
  Interventions: Other: Compounded Pain Cream

INTERVENTIONS:
Other: Compounded Pain Cream — All patients will have been prescribed a topical pain cream prepared by a qualified compounding pharmacy

SUMMARY:
A two-year + 3 Mo. observational study to track compliance and outcomes in adult patients prescribed compounded pharmaceutical creams for the treatment of pain. The project is designed to accumulate tracking information from both patients and physicians over the course of therapy as a supplement to the ordinary care that the patients will normally receive. We seek to discover aspects of successful and unsuccessful treatment using topical pain creams. This information will be analyzed and reports prepared of observations and emergent findings. These reports will be sent during the study every 1 or 2 months to patients, physicians and pharmacists who are participating in the Study. A final compilation of findings and observations will be circulated to participating patients, physicians and pharmacists.

DETAILED DESCRIPTION:
Description Of Data Relevant to Objectives:

The primary objective of this study is to document clinical experience. Specifically, the study will collect:

1. The expectations from both patient and physician. These underlie patient willingness to use a topical therapy, and the physician's motivation in prescribing.
2. What is prescribed and used. The composition of compounded creams vary. Is there an association between the agents / concentrations and the effects on different types of pain?
3. Patterns of use of the creams. Do patients follow the prescription; do they adapt frequency and location of application? Why?
4. What happens with use? Do pain scores change? How quickly, and in what ways do pain scores change with different diagnoses? What is the impact on patient lives? Are expectations typically fulfilled and/or are there surprises and emergent findings?
5. Observations and structured assessments to tabulate the aspects of successful and unsuccessful treatment using topical pain creams of various compositions and for diverse underlying complaints.
6. The level of satisfaction and perceived benefit. If treatment is discontinued, is it because the problem has been resolved? Or is there burden, cost or lack of benefit?
7. Separate confidential information from patients and physicians so that the study team can learn how closely the patients' observations match those of the physicians. The level and nature of the correspondence between patient observations and clinician observations (or lack of it) will be shared in reports sent to study participants. Such reports will not disclose the identities of either physicians or patients.
8. Comments on reports. An area of interest for the study is to investigate the interest in physicians and patients in the reports to be generated concerning the observations from other patients and other physicians. Will patients be interested in their trajectory of treatment? Will sharing the information impact the perceived value of treatment?

Registry Procedures:

1. Data capture is done at visits using structured forms developed in consultation with treating physicians.
2. Patient data: Patients enter ratings and information using encoded paper forms that are then sent by mail directly to the Lexington data entry service, or online using a secure login to send forms to the study database. Such direct from patient transfer is intended to reduce bias that would otherwise influence self assessments of treatment benefit because of the desire of the patient to please the treating physician.
3. Diagnostic standards: International Statistical Classification of Diseases and Related Health Problems, Ninth Revision (ICD9) or International Statistical Classification of Diseases and Related Health Problems, Tenth Revision ( ICD10) codes for diagnosis of pain conditions to be treated are required.
4. Checklists for each visit are completed as part of the trial record to ensure standard processes are followed by treating physicians.
5. If missing or illegible data are not resolvable, then there will be NO imputation. Reports and analysis will be based only on entries where source values were clear. Data entry forms include range and completeness checks, prevention of illogical entry. Free text fields are important for capturing unexpected events and observations. These will be recorded verbatim into the database.
6. There is no primary hypothesis under test. Observations reported will include counts for instances and trends. Assessments and ratings will be reported as averages and distributions.

ELIGIBILITY:
Inclusion Criteria:

* be informed of the nature of the study and must give written informed consent
* be able to communicate effectively with study personnel
* be diagnosed with a condition for which the physician has prescribed a compounded pain cream.

Exclusion Criteria:

* History of allergy or adverse reaction to pain cream ingredients
* History of psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females at least 18 years of age residing in the United States
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in patient reported pain levels following treatment | One year following first patient enrolled
  Across active subjects who have a Baseline pain level AND a followup pain level as of 1 year following first patient enrolled (FPI). Applies to the intended use of the pain cream as established by the diagnosis and area to be treated.

SECONDARY OUTCOMES:
Patient global impression of benefit | One year after first patient enrolled
  Assessed by a structured VAS for completion at followup and final visits. Will be assessed for all patients who have reported on the first followup visit. Mean and distribution will be reported.

OTHER OUTCOMES:
Frequency that patients do NOT use the pain cream as instructed | One year following first patient enrolled (FPI).
  Both incidence (a count and percentage) and 5 most common reasons given by patients for not following the prescription will be reported. The information is proactively captured at followup visits. Baseline establishes prescribed use. Followup items probe for uses inconsistent with prescription. The population will include all subjects as of 1 year following FPI who have reported a followup visit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Raymond, PhD, Study Director — Research and Marketing Consultants
Locations (2):
- United States (2):
  - Lido Chen, Laguna Hills, California
  - Adolphus Anekwe, Gary, Indiana